CLINICAL TRIAL: NCT07304895
Title: Center M Randomized Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: John & Tami Marick Foundation (Unknown)
Responsible Party: Principal Investigator, Ellen Tilden, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00029027
Record Dates: First submitted 2025-12-01; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Perinatal Depression
Keywords: mindfulness based cognitive therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into the Center M intervention or Treatment as Usual (TAU)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be masked to the PI, Co-I's, consultants, and anyone directly collecting or analyzing study data. Primary prenatal care providers will also be masked to subject assignment. Participant and interventionist masking is not possible due to the nature of the intervention arm. The research coordinator(s), research assistants needing to communicate with research participants about group activities (e.g., responding to logistical emails), and volunteers who support the research coordinator or research assistants with communications regarding groups will also be unmasked. Participants will be randomized by the research coordinator or designated research assistant after eligibility determination and study consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Center M (Experimental): In addition to standard prenatal care, participants will participate in Center M sessions, which are weekly one-hour digital group sessions led by a therapist. Each group will include 3-6 participants. The Center M session structure aligns with mindfulness-based cognitive therapy by including mental well-being, core mindfulness and cognitive behavioral therapy skills, in-session practice of skills, and home practice skills. Center M content teaches skills that increase capability for effectively navigating general life stress and the unique stresses of pregnancy and parenting.
  Interventions: Behavioral: Center M
- Treatment as Usual (TAU) (No Intervention): Those randomized to TAU will receive prenatal care as it is standardly delivered in their provider's clinical setting, including perinatal screenings and related educational handouts. Participants will be able to engage in any services recommended by their primary prenatal provider or that they voluntarily initiate, including mental health treatment. Participants will not be proscribed from engaging in other recommended interventions or care.

INTERVENTIONS:
Behavioral: Center M — In addition to standard prenatal care, participants will participate in Center M sessions, which are weekly one-hour digital group sessions led by a therapist. Each group will include 3-6 participants. The Center M session structure aligns with mindfulness-based cognitive therapy by including mental well-being, core mindfulness and cognitive behavioral therapy skills, in-session practice of skills, and home practice skills. Center M content teaches skills that increase capability for effectively navigating general life stress and the unique stresses of pregnancy and parenting.
  Other Names: Mindfulness Based Cognitive Therapy - Perinatal Depression
  Arms: Center M

SUMMARY:
This is a randomized controlled trial with an intervention of Center M compared to treatment as usual. Center M consists of weekly digital one-hour group sessions led by a trained therapist aligned with mindfulness based cognitive therapy. Changes in perinatal depression symptoms will be compared between groups.

DETAILED DESCRIPTION:
The study is a randomized control trial (RCT) with two parallel arms, 1) an intervention arm: Center M added to treatment as usual (TAU), defined as standard prenatal care, and 2) a control arm: TAU, again defined as standard prenatal care. As both groups will be obtaining services through the Center for Women's Health at OHSU, offered standard prenatal care is expected to be similar in both arms. The study will be masked to the PI, Co-I's, consultants, and anyone directly collecting or analyzing study data. Primary prenatal care providers will also be masked to subject assignment. Participant and interventionist masking is not possible due to the nature of the intervention arm. The research coordinator(s), research assistants needing to communicate with research participants about group activities (e.g., responding to logistical emails), and volunteers who support the research coordinator or research assistants with communications regarding groups will also be unmasked. Participants will be randomized by the research coordinator or designated research assistant after eligibility determination and study consent.

The Center M intervention proceeds sequentially with weekly one-hour group sessions led by a trained, masters-level (or equivalent) therapist. Each group will include 3-6 participants. These sessions are conducted digitally via WebEx. Center M session structure aligns with mindfulness based cognitive therapy by including: 1) introduction of a core theme and rationale for how this theme relates to mental well-being (i.e., psychoeducation); 2) teaching core mindfulness (including an emphasis on self-compassion) and CBT skills; 3) facilitating in-session practice of skills (i.e., experiential learning); and 4) reviewing home practice of skills as well as barriers to practice. Sessions are focused on skill development, both through active engagement in practice during group sessions and individual home practice. Center M content teaches skills that increase capability for effectively navigating general life stress and the unique stresses of pregnancy and parenting. It is further designed to increase awareness of early warning signs of perinatal depression to allow for identification of the need for additional resources (including more intensive preventive intervention). The curriculum is designed to be a 'light touch', or minimum necessary intervention that still retains the capacity to prevent perinatal depression. Examples and summaries of the curriculum and accompanying handouts and homework are outlined below and full curriculum, handouts, and homework are available in the IRB documents. The Center M curriculum, handouts and homework follows the parent model MBCT curriculum, with alterations made in direct communication with Sona Dimidjian, PhD, and Sherryl Goodman, PhD, the developers of the parent model. The Center M adaptation has been accomplished with the support and involvement of Drs. Dimidjian and Goodman.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant at ≥ 12 weeks of gestation age (GA)
* ≤ 34 weeks GA at time of Center M intervention initiation
* Receiving prenatal care through the Center for Women's Health at Oregon Health & Science University
* Able to fluently understand, speak and read English
* Available, able and willing to attend online group sessions
* Willing and able to receive home practice materials on an accessible smartphone, tablet or computer
* Residing in Oregon or Washington
* Willingness to participate in either randomization arm

Exclusion Criteria:

* Current or past enrollment in a formal mindfulness-based intervention group
* Score in the "severe" range on the Edinburgh Postnatal Depression Scale (EPDS) (≥ 20) or Patient History Questionnaire (PHQ-9) (≥ 20)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in EPDS scores (baseline to 6 weeks) | Difference between baseline and 6 weeks postpartum
  Measured by the Edinburgh Postnatal Depression Scale (EPDS). EPDS is scored on a scale from 0 to 30 with higher scores representing more symptoms of depression.
Change in PHQ scores (baseline to 6 weeks) | Difference between baseline and 6 weeks postpartum
  Measured by the Patient Health Questionnaire (PHQ-9). PHQ-9 is scored on a scale from 0 to 27 with higher scores representing more symptoms of depression.

SECONDARY OUTCOMES:
Change in EPDS scores (baseline to 3 months) | Difference between baseline and 3 months postpartum
  Measured by the Edinburgh Postnatal Depression Scale (EPDS). EPDS is scored on a scale from 0 to 30 with higher scores representing more symptoms of depression.
Change in PHQ scores (baseline to 3 months) | Difference between baseline and 3 months postpartum
  Measured by the Patient Health Questionnaire (PHQ-9). PHQ-9 is scored on a scale from 0 to 27 with higher scores representing more symptoms of depression.
Change in Mindfulness | Compared between baseline and following the 4 week intervention, between 30 and 38 weeks of gestation.
  Measured by the Five Facet Mindfulness Questionnaire (FFMQ). Average total score can be between 1 and 5 with 5 representing the highest level of mindfulness.
Change in Emotional Regulation | Compared between baseline and following the 4 week intervention, between 30 and 38 weeks of gestation.
  Measured by the Emotional Regulation Questionnaire (ERQ). It consists of two subscales, reappraisal and suppression. For the reappraisal subscale, scores can be between 6 and 42 with higher scores representing a more positive outcome. For the suppression subscale, scores can be between 4 and 28 with a higher score representing a worse outcome.